CLINICAL TRIAL: NCT04115371
Title: A Randomized Controlled Trial of Geriatric Emergency Department Innovations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Scott Dresden, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01HS026489 (AHRQ)
Record Dates: First submitted 2019-09-30; First posted 2019-10-04 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard emergency department care
- Intervention (Other): Standard emergency department are plus GEDI consult
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Geriatric assessment and care coordination provided by a multidisciplinary team in the emergency department including transitional care nurses, social workers, pharmacists, occupational therapists, and physical therapists.
  Arms: Intervention

SUMMARY:
This study evaluates the Geriatric Emergency Department Innovations (GEDI) program at Northwestern Memorial Hospital to care for older adults in the emergency department. Half of the patients will be cared for by a standard ED team plus the GEDI team, while half of the patients will receive usual ED care.

DETAILED DESCRIPTION:
Hospitalization is common for older adults in the Emergency Department (ED) but it carries significant risks including the development of delirium, falls, and nosocomial infections. The Geriatric Emergency Department Innovations (GEDI) program at Northwestern Memorial Hospital attempts to identify and address health related risks for older adults without exposing them to the risks of hospitalization,. GEDI is a unique program consisting of a multidisciplinary team of Transitional Care Nurses (TCN), social workers, pharmacists, occupational therapists and physical therapists who perform ED-based geriatric assessment and care coordination.

To determine the impact of GEDI on health services use and Health Related Quality-of-Life (HRQoL) we will conduct a randomized controlled trial comparing GEDI compared to usual ED care(which often involves hospitalization).

ELIGIBILITY:
Inclusion Criteria:

Northwestern Emergency Department patients who are:

* 65 years or older
* living independently or with friends, family, or caregivers in the community
* Clinical Frailty Scale (CFS) score of 4 or greater

Exclusion Criteria:

Patients will be excluded if they:

* Tested positive for COVID-19
* Are unable to complete the assessments in English
* Are unable to provide informed consent with no Legally Authorized Representative Present or are unable to complete follow-up participation
* Are held in the ED involuntarily as a prisoner or patient with a psychiatric complaint
* Are enrolled in another study to avoid patient fatigue and confounding
* Received a GEDI, Social Work, Pharmacy, or Physical Therapy consult outside of this trial during the current ED visit
* Leave the ED against medical advice or without being seen by a physician
* Are admitted to the ICU
* Are too medically unstable to participate in the assessment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 822 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with hospital admission or death | 30 days
  A composite measure of any hospitalizations or death during the index ED visit or within the follow up time frame

SECONDARY OUTCOMES:
PROMIS-Preference | 9 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS)-Preference (PROPr) score summarizes multiple domains into a single score anchored at 0 (as bad as dead) and 1 (perfect or ideal health). This score quantifies the value that individuals place on different states of health. Preference-based scores can be used in cost-utility analyses and to estimate quality-adjusted life years (QALYs).
  PROPr is calculated from the scores for the 7 PROMIS domains: Cognition, Depression, Fatigue, Pain Interference, Physical Function, Sleep Disturbance, and Ability to Participate in Social Roles and Activities.
  Preference-based scores PROMIS domain scores can be calculated using the HealthMeasures Scoring Service. The HealthMeasures Scoring Service export includes PROMIS theta values used to calculate PROPr using Multi-Attribute Utility Theory (MAUT) which is available at https://github.com/janelhanmer/PROPr
PROMIS-Preference | 30 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS)-Preference (PROPr) score summarizes multiple domains into a single score anchored at 0 (as bad as dead) and 1 (perfect or ideal health). This score quantifies the value that individuals place on different states of health. Preference-based scores can be used in cost-utility analyses and to estimate quality-adjusted life years (QALYs).
  PROPr is calculated from the scores for the 7 PROMIS domains: Cognition, Depression, Fatigue, Pain Interference, Physical Function, Sleep Disturbance, and Ability to Participate in Social Roles and Activities.
  Preference-based scores PROMIS domain scores can be calculated using the HealthMeasures Scoring Service. The HealthMeasures Scoring Service export includes PROMIS theta values used to calculate PROPr using Multi-Attribute Utility Theory (MAUT) which is available at https://github.com/janelhanmer/PROPr
Return Emergency Department Visits | 9 days
  Any Emergency Department Visits which occurs after the ED encounter in which the patient was enrolled in the study.
Return Emergency Department Visits | 30 days
  Any Emergency Department Visits which occurs after the ED encounter in which the patient was enrolled in the study.
Death | 9 days
  All cause death
Death | 30 days
  All cause death
PROMIS Item Bank v2.0 - Physical Function (Adaptive) | 9 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Item Bank uses Computer Adaptive Testing (CAT) in which participant responses guide the system's choice of subsequent items from the full item bank (165 items in total in adult bank). Although items differ across respondents taking CAT, scores are comparable across participants.
  Measure Description: PROMIS subscale for physical function assesses the extent to which patients' perceived capability rather than actual performance of physical activities using a 5-point Likert scale. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. T-scores range from 20 to 80. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Item Bank v2.0 - Physical Function (Adaptive) | 30 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Item Bank uses Computer Adaptive Testing (CAT) in which participant responses guide the system's choice of subsequent items from the full item bank (165 items in total in adult bank). Although items differ across respondents taking CAT, scores are comparable across participants.
  Measure Description: PROMIS subscale for physical function assesses the extent to which patients' perceived capability rather than actual performance of physical activities using a 5-point Likert scale. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. T-scores range from 20 to 80. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Item Bank v2.0 - Ability to Participate Social Roles and Activities (Adaptive) | 9 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities Item Bank uses Computer Adaptive Testing (CAT) in which participant responses guide the system's choice of subsequent items from the full item bank (35 items in total). Although items differ across respondents taking CAT, scores are comparable across participants.
  Measure Description: PROMIS item bank for ability to participate in social roles and activities assesses the extent to which patients' perceived ability to perform one's usual social roles and activities using a 5-point Likert scale. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. T-scores range from 20 to 80. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Item Bank v2.0 - Ability to Participate Social (Adaptive) | 30 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities Item Bank uses Computer Adaptive Testing (CAT) in which participant responses guide the system's choice of subsequent items from the full item bank (35 items in total). Although items differ across respondents taking CAT, scores are comparable across participants.
  Measure Description: PROMIS item bank for ability to participate in social roles and activities assesses the extent to which patients' perceived ability to perform one's usual social roles and activities using a 5-point Likert scale. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. T-scores range from 20 to 80. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Item Bank v. 1.0 - Emotional Distress - Anxiety (Adaptive) | 9 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Item Bank uses Computer Adaptive Testing (CAT) in which participant responses guide the system's choice of subsequent items from the full item bank (29 items in total). Although items differ across respondents taking CAT, scores are comparable across participants.
  Measure Description: PROMIS item bank for anxiety assesses the extent to which patients experience anxiety symptoms over the past 7 days using a 5-point Likert scale. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. T-scores range from 20 to 80. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Item Bank v. 1.0 - Emotional Distress - Anxiety (Adaptive) | 30 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Item Bank uses Computer Adaptive Testing (CAT) in which participant responses guide the system's choice of subsequent items from the full item bank (29 items in total). Although items differ across respondents taking CAT, scores are comparable across participants.
  Measure Description: PROMIS item bank for anxiety assesses the extent to which patients experience anxiety symptoms over the past 7 days using a 5-point Likert scale. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. T-scores range from 20 to 80. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Item Bank v. 1.0 - Emotional Distress - Depression (Adaptive) | 9 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Item Bank uses Computer Adaptive Testing (CAT) in which participant responses guide the system's choice of subsequent items from the full item bank (28 items in total). Although items differ across respondents taking CAT, scores are comparable across participants.
  Measure Description: PROMIS item bank for depression assesses the extent to which patients experience depressive symptoms over the past 7 days using a 5-point Likert scale. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. T-scores range from 20 to 80. A higher PROMIS T-score represents more of the concept being measured.
PROMIS Item Bank v. 1.0 - Emotional Distress - Depression (Adaptive) | 30 days
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Item Bank uses Computer Adaptive Testing (CAT) in which participant responses guide the system's choice of subsequent items from the full item bank (28 items in total). Although items differ across respondents taking CAT, scores are comparable across participants.
  Measure Description: PROMIS item bank for depression assesses the extent to which patients experience depressive symptoms over the past 7 days using a 5-point Likert scale. PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. T-scores range from 20 to 80. A higher PROMIS T-score represents more of the concept being measured.
Number of patients admitted | 24 hours
  A patient who is admitted to inpatient status during the emergency department visit in which they are enrolled in the study
Number of patients admitted | 9 days
  A patient who is admitted to inpatient status during the emergency department visit in which they are enrolled in the study or within the follow up time frame
Number of patients admitted | 30 days
  A patient who is admitted to inpatient status during the emergency department visit in which they are enrolled in the study or within the follow up time frame
Number of patients with hospital admission or death | 9 days
  A composite measure of any hospitalizations or death during the index ED visit or within the follow up time frame

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Dresden, MD, MS, Principal Investigator — Northwestern University Department of Emergency Medicine
Locations (1):
- Northwestern University Department of Emergency Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The Galter Library at Northwestern University has implemented a DigitalHub to facilitate the storage and sharing of research products, including data sets, presentations, documentation, brochures, etc. The DigitalHub also provides digital object identifier so that these resources can be appropriately cited and tracked.
  Where feasible we will curate and make available structured data both as de-identified and limited datasets as defined under HIPAA.
  Interested collaborators will complete an online collaborative research request survey.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available at the completion of the study and will be available for at least 5 years.
Access Criteria: Access will be determined by the DigitalHub requirements.
URL: https://digitalhub.northwestern.edu/

REFERENCES:
- [Derived] Dresden SM, Lo AX, Lindquist LA, Kocherginsky M, Post LA, French DD, Gray E, Heinemann AW. The impact of Geriatric Emergency Department Innovations (GEDI) on health services use, health related quality of life, and costs: Protocol for a randomized controlled trial. Contemp Clin Trials. 2020 Oct;97:106125. doi: 10.1016/j.cct.2020.106125. Epub 2020 Aug 26. PMID 32858227